CLINICAL TRIAL: NCT01410903
Title: Immunoadsorption in Addition to the Established Therapy in Patients With Systemic Sclerosis
Brief Title: Immunoadsorption in Patients With Severe Systemic Sclerosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inadequately recruitment rate, funding is not secured
Sponsor: GWT-TUD GmbH (Other)
Collaborators: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IAS - SSc 2010
Record Dates: First submitted 2011-08-04; First posted 2011-08-05 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Systemic Scleroderma
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TheraSorb Ig (Experimental)
  Interventions: Device: TheraSorb Ig

INTERVENTIONS:
Device: TheraSorb Ig — 1,5 plasma volume per treatment venovenous immunoadsorption frequency: three times weekly in week 1 and 2, two times weekly in week 3-6, two times two-weekly in week 7-12 duration: 12 months
  Other Names: Ig-TheraSorb; code 330-000-452

SUMMARY:
The purpose of this study is to evaluate source data for the survival and the investigation of the preliminary efficacy of immunoadsorption in patients with severe systemic sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* systemic sclerosis according to the ACE-criteria
* severe pulmonary manifestation with reduced DLCO
* signed informed consent

Exclusion Criteria:

* inadequate peripheral venous access
* participation in another clinical trial
* heart failure
* pronounced allergic diathesis, particularly in case of known hypersensitivity to drugs and/or materials used in the extracorporeal circuit

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
survival under immunoadsorption | 6 months

SECONDARY OUTCOMES:
survival under immunoadsorption | 12 months
Number of Serious Adverse Events | 12 months
change in "modified Rodnan Skin Score" | 12 months
change in Diffusing Capacity of the Lung for Carbon Monoxide | 12 months
change in Scleroderma Health Assenssment Questionnaire | 12 months
change of pulmonary arterial pressure | 12 months
reoccurrence of finger ulcers | 12 months
healing of finger ulcers | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin Aringer, Prof., Principal Investigator — Universitätsklinikum Dresden
Locations (1):
- Universitätsklinikum Dresden, Dresden, Germany